CLINICAL TRIAL: NCT05872230
Title: Massage Percussion Therapy for Passage of Urolithiasis Fragments After Ureteroscopy
Brief Title: Massage Percussion for Passage of Urolithiasis Fragments After Ureteroscopy.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigators terminated study given recent advancements in ureteroscopic technique and suction technique.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Ryan Hsi, Urologist, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VUMC01
Record Dates: First submitted 2023-05-04; First posted 2023-05-24 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Nephrolithiasis
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control (No Intervention): Patient receives standard postoperative care with no percussion therapy.
- PACU percussion (Experimental): Patient receives percussion therapy in the PACU immediately after surgery.
  Interventions: Device: Massage Percussion Therapy device
- Postoperative appointment percussion (Experimental): Patient receives percussion therapy in the office on the day of follow up.
  Interventions: Device: Massage Percussion Therapy device
- Both PACU and Postop appointment percussion. (Experimental): Patient receives percussion therapy in the PACU and receives percussion therapy in the office on the day of follow up.
  Interventions: Device: Massage Percussion Therapy device

INTERVENTIONS:
Device: Massage Percussion Therapy device — Using massage percussion postoperatively.
  Arms: Both PACU and Postop appointment percussion.; PACU percussion; Postoperative appointment percussion

SUMMARY:
Flexible ureteroscopy is characterized as first-line therapy for renal stones < 2 cm in size. Stones are commonly treated with dusting or fragmentation techniques which requires passage of stone fragments after surgery. Quoted stone free rate after flexible ureteroscopy is approximately 40-60% with a dusting technique. Residual fragments are often under 1mm in size and can layer in the lower pole of the kidney, complicating spontaneous stone passage. Improving the stone free rate after surgery decreases the need for secondary surgeries and decreases risk of future stone events.

Numerous techniques have been proposed to increase stone passage including positional changes and percussion therapy. To date, there is overall limited data a lack of techniques that can be readily available in the outpatient setting, easily added to scheduled appointments, reproducible results and well tolerated by patients.

DETAILED DESCRIPTION:
Researchers in China have developed a proprietary oscillation machine to be used in an outpatient setting. The External Physical Vibration Lithecbole (EPVL) is used to provide vibration after stone fragmentation to facilitate movement of fragments into a more favorable orientation for stone passage. After extracorporeal shockwave lithotripsy and ureteroscopy, use of EPVL after surgery has been shown to increase stone free rate.

Chest percussion for cystic fibrosis patients has been adapted for use after ureteroscopy. After undergoing extracorporeal shockwave lithotripsy, patients are placed in a percussion physiotherapy vest, given diuretics and positioned in Trendelenburg. Imaging obtained before and after percussion demonstrates successful stone movement and increases stone free rates in several different protocols compared to patients who do not receive percussive therapy.

Percussion therapy is clearly effective to improve stone free rates after ureteroscopy and is effective regardless of technique, protocol, or percussive device. However, proposed techniques with EPVL and chest physiotherapy vests can be expensive, cumbersome and require specialty equipment. In addition, proposed equipment in prior studies is not readily available in outpatient clinics.

ELIGIBILITY:
Inclusion Criteria:

* Any patient after treatment of renal stones with ureteroscopy during which residual stone fragments (less than 2mm by surgeon estimation) is left in the kidney.
* Must be 18 years or older
* Must be able to give consent
* Preoperative abdominal CT

Exclusion Criteria:

* On pharmacologic anticoagulation. Aspirin up to 81mg will be allowed.
* Cannot tolerate flank, prone or Trendelenburg position.
* Cannot tolerate percussion.
* History of acute rib fractures or osteopenia/osteoporosis.
* Any patient who is on a fluid intake restriction.
* Pregnancy
* Untreated UTI
* History of struvite stones
* Requiring a planned secondary stone procedure within 90 days
* If stent must stay in longer than 10 days
* Ureteral stones (without renal stones)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Patients who are able to tolerate and complete the percussion therapy. | Postop day 0-10.
  If patients can tolerate the percussion therapy in the treatment arms. This is evaluated by patients being able to complete the percussion therapy session and completing pain questionnaires.
Stone Free Rate. | 6 weeks after surgery.
  Patients will have standard postoperative imaging at six weeks, as is standard of care. Presence of stone fragments and fragment size will determine the postoperative stone free rate.

SECONDARY OUTCOMES:
weight of passed stone fragments | 6 weeks.
  PAtients will strain urine to collect stone fragments after surgery until stent removal. The stone fragments will be sent for stone analysis, as is standard of care, during which fragments will be weighed.
Unplanned return visits. | 6 weeks.
  Follow patients who have unplanned return trips to the ED or the clinic for pain or complications after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Hsi, Principal Investigator — VUMC
Locations (1):
- University of Montreal, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No